CLINICAL TRIAL: NCT04379973
Title: Live Birth After Additional Tubal Flushing With Oil-based Contrast Versus no Additional Flushing: a Randomised, Multicentre, Parallel Group Pragmatic Trial in Infertile Women With at Least One Patent Tube at Hysterosalpingo-foam Sonography
Brief Title: Live Birth After Additional Tubal Flushing With Oil-based Contrast Versus no Additional Flushing:
Acronym: HYFOIL
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dafne Balemans (Other)
Responsible Party: Sponsor-Investigator, Dafne Balemans, Clinical Trial Center, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYOIL
Record Dates: First submitted 2020-04-23; First posted 2020-05-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubal flush with Lipiodol Ultra Fluide® after Hyfosy (Experimental)
  Interventions: Drug: Lipiodol Ultra Fluide®
- No tubal flush after Hyfosy (No Intervention)

INTERVENTIONS:
Drug: Lipiodol Ultra Fluide® — Tubal flush with 5-10mL oil-soluble contrast medium (OSCM) (Lipiodol Ultra Fluide®, Guerbet, France) immediately after Hyfosy. The use will be off-label.
  Arms: Tubal flush with Lipiodol Ultra Fluide® after Hyfosy

SUMMARY:
Ten to 15 percent of couples in their reproductive lifetime face fertility problems which is defined by WHO as the absence of pregnancy after minimal 12 months of unprotected sexual intercourse. The three most frequent causes of subfertility are: sperm defects, ovulation disorders and tubal pathology. In order to exclude tubal pathology, tubal patency tests are performed under ultrasound guidance with foam (hysterosalpingo-foam sonography (Hyfosy)) or with contrast/water (hysterosalpingo-contrast sonography (Hycosy)).

This trial will investigate whether tubal flushing with an oil-soluble contrast medium (OSCM) can increase the likelihood of a spontaneous conception after tubal patency testing with Hyfosy under ultrasound guidance compared to no additional flushing in a population of infertile women between 18 and 40 years of age with absence of pregnancy after 12 months of unprotected sexual intercourse or who have three cycles of donor insemination without pregnancy or three ovulatory ovulation induction cycles without pregnancy. The use of Lipiodol Ultra Fluide® is off-label in Hyfosy.

This multicenter, randomised, open-label, comparative and pragmatic trial compares 2 arms which will be randomised 1:1:

* Intervention group: Tubal flush with 5-10mL oil-soluble contrast medium (Lipiodol Ultra Fluide®, Guerbet, France) immediately after Hyfosy
* Control group: No additional intervention after Hyfosy The study comprises a screening period of maximum 8 weeks (w-8 to d1), randomisation (w-8 to d1), a start study visit at which the Hyfosy is performed (d1) and a fertility treatment period of 6 months (d1-w26). If the woman is not pregnant at 6 months after Hyfosy, the follow-up will last till 12 months (w52). If the participant is pregnant at 6 months after Hyfosy, the follow-up will last till maximal 4 months after live birth or miscarriage.

The primary endpoint is the occurrence of live birth, with the first day of the last menstrual cycle in which the patient conceives within 6 months after Hyfosy. Secondary endpoints consist of reproductive outcomes, gestational age at delivery, birth weight, neonatal mortality, major congenital anomaly, neonatal outcomes and thyroid function, pregnancy complications, number of complications during or immediately after the intervention, pain score of the Hyfosy and additional flush, thyroid function of the mother, general and disease-specific quality of life.

ELIGIBILITY:
Inclusion Criteria:

Infertile women undergoing Hyfosy as part of the fertility workup. Women will be eligible if they

* are ≥ 18 years and < 40 years
* have infertility defined as

  * lack of conception despite 12 months of unprotected intercourse OR;
  * if they are taking part in a donor sperm insemination programme: three cycles of donor insemination without pregnancy OR;
  * in case of treated ovulation disorder: three ovulatory ovulation induction cycles without pregnancy
* have tubal patency of at least one Fallopian tube on Hyfosy

Exclusion Criteria:

Women with

* known iodine allergy
* allergy to poppy seed oil
* ovulation disorders defined as less than eight menstrual cycles per year who did not have three ovulatory cycles after ovulation induction
* contra-indication to have tubal patency testing according to the site's indication
* active thyroid disorders
* untreated subclinical hypothyroidism (TSH>2.5mIU/L) in case of auto-immune thyroid disease
* uterine surgery in the past two months before Hyfosy
* a male partner (if applicable)

  * with a post-wash Total Motile Sperm Count (TMC) < 1x106 and/or TMC < 3x106 in the native sperm analysis [TMC is defined as volume X concentration X (A* (progressive) + B* (non progressive) motility in %) divided by 100] OR
  * with a history suspect of severe male factor infertility if no sperm sample is available at time of randomisation
* an indication for IVF defined as patients who are advised to go to IVF immediately because of bilateral tubal block, severe male factor infertility, unsolved anovulatory problems, endometriosis with residual functional problems"
* no Belgian national number (RRN/INS)

  * A+B when A,B,C is used (WHO 2010) A+B+C when A,B,C, D is used (WHO 2021)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 736 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Live birth | Delivery
  the occurrence of live birth, counting from the first day of the last menstrual cycle in which the patient conceives within 6 months after Hyfosy.

SECONDARY OUTCOMES:
Type of pregnancy | 15 months after Hyfosy
  single or multiple pregnancy
Number of miscarriages | 15 months after Hyfosy
  presence of miscarriages
Amount of pregnancy complications | 15 months after Hyfosy
  gestational diabetes, hypertensive disease, placenta praevia, intrauterin growth restriction, premature birth
Number of ectopic pregnancies | 15 months after Hyfosy
  the presence of ectopic pregnancy
Number of clinical pregnancies | 15 months after Hyfosy
  the presence of clinical pregnancy
Complication during or after Hyfosy with intervention | immediately after intervention
  embolism, anaphylactic shock, pelvic inflammatory disease, intravasation, infection and hemorrhage
Pain score of the Hyfosy with or without intervention | immediately after Hyfosy
  VAS (0 = no pain; 10 = worst possible pain)
Pain score of the intervention with IMP if applicable | immediately after intervention
  VAS (0 = no pain; 10 = worst possible pain)
Thyroid function of baby | 3 days after delivery
  heel prick test (TSH, FT4)
Birthweight | at delivery
  Birthweight of baby
Gestational age at delivery | at delivery
  Live birth after how many weeks pregnancy
Neonatal care | at delivery
  Neonatal care (Yes/No)
Number of babies | at delivery
  Number of babies after live birth
Maternal thyroid function | 4 weeks, 26 weeks, 15 weeks after delivery
  TSH, FT4 determination
General quality of life | 26 weeks
  EuroQol-5D-5Levels (EQ-5D-5L):
  Level 1: indicating no problem Level 2: indicating slightproblems Level 3: indicating moderateproblems Level 4: indicating severe problems Level 5:indicating extreme problems; VAS (score 0 = worst health status; score 100 = best health status) How higher the score, how better the quality of life
Disease-specific quality of life | 26 weeks
  Fertility Quality Of Life tool (FertiQol):
  1. Very poor (0), poor (1), neither poor nor good (2), very good (4)
  2. Very dissatisfied (0), dissatisfied (1), neither satisfied nor dissatisfied (2), satisfied (3), very satisfied (4)
  3. Always (0), very often (1), quite often (2), Seldom (3), never (4)
  4. An extreme amount (0), very much (1), a moderate amount (2), a little (3), not at all (4)
  5. Completely (0), a great deal (1), moderately (2), not much (3), not at all (4)
  Scores on the response scales are reversed, summed and scaled to range from 0 to 100. Higher scores on the subscales and total scores indicate better quality of life
Neonatal Mortality | at delivery
  Neonatal death after delivery
Major Congenital Anomaly | at delivery
  Neonatal major anomaly
Gender of baby | at delivery
  Gender of baby (M/F)

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (16):
  - Antwerp University Hospital, Antwerp
  - GZA Sint Augustinus, Antwerp
  - Imelda, Bonheiden
  - AZ Klina, Brasschaat
  - AZ Sint Jan Brugge, Bruges
  - CHIREC, Brussels
  - UCL Saint Luc, Brussels
  - UZ Brussel, Brussels
  - Ziekenhuis Oost Limburg, Genk
  - AZ Sint Lucas, Ghent
  - UZ Gent, Ghent
  - Hôpital Erasme, Lennik
  - UZ Leuven, Leuven
  - CHC Mont Légia, Liège
  - CHR Citadelle, Liège
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Neubourg D, Janssens L, Verhaegen I, Smits E, Mol BW, Roelant E. Live birth after additional tubal flushing with oil-based contrast versus no additional flushing: a randomised, multicentre, parallel-group pragmatic trial in infertile women with at least one patent tube at hysterosalpingo-foam sonography (HYFOIL study). BMJ Open. 2021 Nov 29;11(11):e054845. doi: 10.1136/bmjopen-2021-054845. PMID 34845077